CLINICAL TRIAL: NCT00723632
Title: Cost of Treatment of Chronic Hepatitis C Using Combination of Peginterferon α-2b Plus Ribavirin
Brief Title: Pharmacoeconomic Study Assessing the Cost of Chronic Hepatitis C Treatment With Peginterferon Alfa-2b (PegIntron) and Ribavirin (Rebetol) in the Czech Republic (Study P04588)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04588
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2011-12-20 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peginterferon alfa-2b and ribavirin: All participants included in the study
  Interventions: Biological: peginterferon alfa-2b; Drug: ribavirin

INTERVENTIONS:
Biological: peginterferon alfa-2b — Peginterferon alfa-2b administered in accordance with approved labeling, ie, 1.5 μg/kg weekly SC for 48 weeks for participants with hepatitis C virus (HCV) genotype 1 or for 24 weeks for participants with HCV genotype 2, 3.
  Other Names: SCH 054031; PegIntron; peginterferon α-2b
Drug: ribavirin — Ribavirin administered in accordance with approved labeling, ie, 800 mg/day for participants <65 kg, 1000 mg/day for participants >65 to <85 kg, and 1200 mg/day for participants >=85 kg, administered orally for 48 weeks for participants with HCV genotype 1 or for 24 weeks for participants with HCV genotype 2, 3.
  Other Names: SCH 018908; Rebetol

SUMMARY:
The objective of the study is to evaluate the costs associated with peginterferon alfa-2b (PegIntron) plus ribavirin (Rebetol) treatment for chronic hepatitis C in the Czech Republic. Only costs associated with rescue medication, concomitant therapy, disease monitoring, and medical intervention costs recognized by the treating institution as treatment-related expenses will be included in the analysis. The study will also evaluate the correlation between hepatitis C virus (HCV) therapy-related costs with ribavirin dosing and participant history.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic hepatitis C
* At least 18 years old
* Eligibility determined based on the diagnosis and medical judgment only.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic hepatitis C treated with peginterferon alfa-2b and ribavirin at approximately 81 sites in the Czech Republic.
Sampling Method: Probability Sample
Enrollment: 901 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon Alfa-2b and Ribavirin: Participants received peginterferon alfa-2b administered subcutaneously 1.5 μg/kg weekly and ribavirin administered orally at 800 mg/day for participants <65 kg, 1000 mg/day for participants >65 to <85 kg, and 1200 mg/day for participants >=85 kg. Treatment was administered for 48 weeks to participants with hepatitis C virus (HCV) genotype 1 or for 24 weeks to participants with HCV genotype 2, 3.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Started | 901
Completed | 698 (Completed initial exam form and >= 1 follow up visit form; end of treatment and SVR status recorded)
Not Completed | 203

BASELINE CHARACTERISTICS:
Groups:
- Peginterferon Alfa-2b and Ribavirin: Participants received peginterferon alfa-2b administered subcutaneously 1.5 μg/kg weekly and ribavirin administered orally at 800 mg/day for participants <65 kg, 1000 mg/day for participants >65 to <85 kg, and 1200 mg/day for participants >=85 kg. Treatment was administered for 48 weeks to participants with HCV genotype 1 or for 24 weeks to participants with HCV genotype 2, 3.
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 698
Age, Continuous [Mean (Full Range); unit: years] — Age is reported for participants in the analysis population
  years | 38 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender is reported for participants in the analysis population
  Participants
    Female | 300
    Male | 398

OUTCOME MEASURES:

1. Primary Outcome: Average Cost Per Participant With Sustained Virologic Response (SVR) Stratified by Weight Category
Description: SVR is defined as undetectable HCV ribonucleic acid (RNA) six months after the end of treatment. Cost per participant with SVR was calculated as a ratio of the total costs for all participants and the number of participants with SVR in the given group. All costs were adjusted for inflation to 2010 values.
Time Frame: From enrollment up to 48 weeks for participants with hepatitis C virus (HCV) genotype 1, and from enrollment up to 24 weeks for participants with HCV genotypes 2 and 3
Population: Participants were included in the analysis if all of the following conditions were met: initial exam form was completed; at least 1 follow up visit form was completed; the end of treatment (either according to plan or early) was recorded; and SVR status was recorded six months after treatment termination.
Measure: Mean (Full Range); unit: Czech Crown
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 698
Czech Crown
  <= 64 kg (n=182) | 28,271 [24,461 to 33,676]
  65-85 kg (n=334) | 31,429 [27,027 to 36,989]
  >= 85 kg (n=182) | 34,782 [29,243 to 42,261]

2. Secondary Outcome: Average Cost Per Participant With SVR Stratified by Ribavirin Dosage
Description: as for outcome 1
Time Frame: From enrollment up to 48 weeks for participants with HCV genotype 1, and from enrollment up to 24 weeks for participants with HCV genotypes 2 and 3
Population: as for outcome 1
Measure: Mean (Full Range); unit: Czech Crown
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 698
Czech Crown
  800 mg/day (n=167) | 31,119 [24,658 to 39,587]
  1000 mg/day (n=333) | 29,306 [26,047 to 33,388]
  1200 mg/day (n=198) | 35,621 [30,233 to 43,274]

3. Secondary Outcome: Average Cost Per Participant With SVR Stratified by Prior Treatment Status
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Full Range); unit: Czech Crown
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 698
Czech Crown
  Treatment-Naive (n=543) | 30,109 [27,180 to 33,580]
  Previously Treated (n=155) | 37,486 [29,938 to 48,682]

ADVERSE EVENTS:
Description: Serious adverse events and non-serious adverse events were not required to be captured as part of the study database, and were reported directly to the Sponsor. Therefore, no adverse events were collected, and the number at risk is zero.
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No